CLINICAL TRIAL: NCT04503603
Title: A Randomized, Double-blind, Placebo-Controlled, Repeat-dose, Single-center Phase 1a Study to Determine the Safety, Tolerability, and Pharmacokinetics of Lanadelumab Administered Intravenously in Healthy Adult Volunteer Subjects
Brief Title: A Study to Determine the Safety, Tolerability, and Pharmacokinetics of Lanadelumab Administered Intravenously in Healthy Adult Volunteer Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-743-1003
Record Dates: First submitted 2020-08-05; First posted 2020-08-07 (Actual); Results first posted 2022-03-07 (Actual); Last update posted 2022-03-07 (Actual); Status verified 2021-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — lanadelumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Lanadelumab 300 mg (Experimental): Participants will receive single dose of lanadelumab 300 mg intravenous (IV) infusion on Day 1 followed by second dose on Day 4.
  Interventions: Drug: Lanadelumab
- Placebo (Placebo Comparator): Participant will receive single dose of lanadelumab matching placebo (normal saline) IV infusion on Day 1 followed by second dose on Day 4.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Lanadelumab — Participants will receive lanadelumab 300 mg IV infusion on Day 1 followed by Day 4.
  Other Names: TAK-743
  Arms: Lanadelumab 300 mg
Other: Placebo — Participants will receive placebo matching to lanadelumab IV infusion on Day 1 followed by Day 4.
  Arms: Placebo

SUMMARY:
The purpose of this study to evaluate the safety, tolerability and pharmacokinetics (PK) of lanadelumab administered by Intravenous (IV) infusion in healthy adult volunteers.

DETAILED DESCRIPTION:
A Randomized, Double-blind, Placebo-Controlled, Repeat-dose, Single-center Phase 1a Study to Determine the Safety, Tolerability, and Pharmacokinetics of Lanadelumab Administered Intravenously in Healthy Adult Volunteer Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 19-55 years of age, inclusive, at screening.
* Continuous non-smoker who has not used nicotine-containing products for at least 30 days prior to the first dosing and throughout the study, based on participant self-reporting.
* Body mass index (BMI) greater than or equal to (>=) 18.0 and less than or equal to (<=) 32.0 kilogram per square meter (kg/m^2) at screening.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, vital signs or electrocardiograms (ECGs), per the investigator.
* Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol or females of non-childbearing potential.
* Understands the study procedures in the informed consent form (ICF) and be willing and able to comply with the protocol.

Exclusion Criteria:

* Is mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
* History or presence of clinically significant medical or psychiatric condition or disease per the investigator.
* History of any illness that might confound the results of the study or poses an additional risk to the participant by their participation in the study, per the investigator.
* History or presence of alcoholism or drug abuse within the past 2 years prior to the first dosing per the investigator.
* History or presence of hypersensitivity or idiosyncratic reaction to the study drug(s) or related compounds.
* History or presence of any hematological, hepatic, respiratory, cardiovascular, renal, neurological or psychiatric disease, gall bladder removal, or current or recurrent disease that could affect the action, absorption, or disposition of the investigational product, or clinically significant clinical or laboratory assessments per the investigator.
* Female participants with a positive pregnancy test or lactating.
* Positive urine drug or alcohol results at screening.
* Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV).
* Supine blood pressure is less than 90/40 millimetre of mercury (mmHg) or greater than 140/90 mmHg at screening.
* Supine heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
* Orthostatic vital sign results with a decrease in systolic greater than (>) 20 mmHg or decrease in diastolic > 10 mmHg and increase in pulse of > 20 beats per minute.
* QTcF interval is > 450 milliseconds (msec) (males) or > 470 msec (females) or ECG findings are deemed abnormal with clinical significance at screening per the investigator.
* Estimated creatinine clearance less than (<) 80 milliliters per minute (mL/min) at screening.
* Unable to refrain from or anticipates the use of any drug, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing and throughout the study. Medication listed as part of acceptable birth control methods will be allowed. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first study drug administration. After randomization/dosing, a nonsteroidal anti-inflammatory drug may be administered at the discretion of the investigator. Hormone replacement therapy will also be allowed if the participant has been on the same stable dose for the immediate 3 months prior to first study drug administration.
* Has been on a diet incompatible with the on-study diet, per the investigator, within the 30 days prior to the first dosing and throughout the study.
* Donation of blood or significant blood loss within 56 days prior to the first dosing.
* Plasma donation within 7 days prior to the first dosing.
* Participation in another clinical study within 30 days or 5 half-lives prior to the first dosing. The 30-day window or 5 half-lives will be derived from the date of the last blood collection or dosing, whichever is later, in the previous study to Day 1 of the current study

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda Development Center Americas, Inc.
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/5f9c5f6a2f8e61001ef3242d

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 1 investigative site in the United States between 10 August 2020 (first participant first visit) and 23 December 2020 (last participant last visit).
Pre-assignment Details: A total of 12 healthy participants were enrolled and randomized to receive lanadelumab 300 milligrams (mg) or matching placebo in this study.
Groups:
- Lanadelumab 300 mg: Participants received a single dose of lanadelumab 300 mg intravenous (IV) infusion on Day 1 followed by a second dose on Day 4.
- Placebo: Participants received a single dose of lanadelumab matching placebo (normal saline) IV infusion on Day 1 followed by a second dose on Day 4.
Period: Overall Study
Arm/Group | Lanadelumab 300 mg | Placebo
Started | 9 | 3
Completed | 9 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set consisted of all participants who had started at least 1 dose of lanadelumab or placebo.
Groups:
- Lanadelumab 300 mg: Participants received a single dose of lanadelumab 300 mg IV infusion on Day 1 followed by a second dose on Day 4.
- Placebo: Participants received a single dose of placebo (normal saline) IV infusion on Day 1 followed by a second dose on Day 4.
- Total: Total of all reporting groups
Arm/Group | Lanadelumab 300 mg | Placebo | Total
Number analyzed (Participants) | 9 | 3 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.3 (11.73) | 42.0 (10.44) | 36.3 (11.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 1 | 5
  Male | 5 | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 9 | 2 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 5 | 3 | 8
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study that did not necessarily have a causal relationship with the treatment. TEAEs were events that occurred on or after the date and time of administration of the first dose of study medication. TEAEs included both serious TEAEs and non-serious TEAEs. Number of participants with TEAEs were reported.
Time Frame: From the first dose of study treatment up to the end of study (Day 112)
Population: The safety analysis set consisted of all participants who had started at least 1 dose of lanadelumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants | 7 | 2

2. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Laboratory Parameters
Description: Clinical laboratory assessment included hematology, clinical chemistry, coagulation, and urinalysis. Any changes in clinical laboratory results that were deemed clinically significant were judged by the investigator. The number of participants with clinically significant change from baseline in laboratory values were reported.
Time Frame: From the first dose of study treatment up to the end of study (Day 112)
Population: The safety analysis set consisted of all participants who had started at least 1 dose of lanadelumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

3. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included blood pressure (systolic and diastolic), heart rate, and body temperature (oral). Any changes in vital signs that were deemed clinically significant were judged by the investigator. The number of participants with clinically significant change from baseline in vital signs were reported.
Time Frame: From the first dose of study treatment up to the end of study (Day 112)
Population: The safety analysis set consisted of all participants who had started at least 1 dose of lanadelumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

4. Primary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Description: 12-lead ECG recordings included rhythm, heart rate (as measured by RR interval), PR interval, QRS duration, and QT interval. Any changes in ECG parameters that were deemed clinically significant were judged by the investigator. The number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported.
Time Frame: From the first dose of study treatment up to the end of study (Day 112)
Population: The safety analysis set consisted of all participants who had started at least 1 dose of lanadelumab or placebo.
Measure: Count of Participants; unit: Participants
Arm/Group | Lanadelumab 300 mg | Placebo
Number analyzed (Participants) | 9 | 3
Participants | 0 | 0

5. Primary Outcome: AUC0-last: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Quantifiable Concentration for Lanadelumab
Description: AUC0-last for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: The pharmacokinetic (PK) analysis set consisted of all participants who received at least one dose of the study drug and had at least one evaluable PK concentration post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hour*microgram per milliliter (h*mcg/mL)
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
hour*microgram per milliliter (h*mcg/mL) | 32955 (10.5)

6. Primary Outcome: AUC0-inf: Area Under the Plasma Concentration-time Curve From Time Zero Extrapolated to Infinity for Lanadelumab
Description: AUC0-inf for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: The PK analysis set consisted of all participants who received at least one dose of the study drug and had at least one evaluable PK concentration post-dose.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mcg/mL
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
h*mcg/mL | 33305 (10.5)

7. Primary Outcome: Cmax1: Maximum Observed Plasma Concentration Following the First IV Dose for Lanadelumab
Description: Cmax1 following the first IV dose for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: microgram per milliliter (mcg/mL)
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
microgram per milliliter (mcg/mL) | 75.6 (16.1)

8. Primary Outcome: Cmax2: Maximum Observed Plasma Concentration Following the Second IV Dose for Lanadelumab
Description: Cmax2 following the second IV dose for lanadelumab was reported.
Time Frame: Pre-dose (Day 4) up to 2592 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
mcg/mL | 120 (20.7)

9. Primary Outcome: Tmax1: Minimum Observed Time to Reach the First Cmax1 for Lanadelumab
Description: Tmax1 following the first IV dose for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
hours | 2.01 [2.00 to 4.01]

10. Primary Outcome: Tmax2: Minimum Observed Time to Reach the Second Cmax2 for Lanadelumab
Description: Tmax2 following the second IV dose for lanadelumab was reported.
Time Frame: Pre-dose (Day 4) up to 2592 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: hours
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
hours | 74.03 [72.92 to 76.02]

11. Primary Outcome: Terminal Half-Life (T1/2) of Lanadelumab in Plasma
Description: T1/2 is defined as the time required for the concentration of the drug to reach half of its original value. T1/2 for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: as for outcome 6
Measure: Median (Full Range); unit: days
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
days | 19.3 [13.7 to 19.6]

12. Primary Outcome: Clearance (CL) of Lanadelumab in Plasma
Description: Clearance is defined as a quantitative measure of the rate at which a drug substance is removed from the body. CL for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter per hour (mL/h)
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
milliliter per hour (mL/h) | 18.1 (10.4)

13. Primary Outcome: Vss: Volume of Distribution at Steady State in Plasma for Lanadelumab
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vss for lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milliliter (mL)
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
milliliter (mL) | 8070 (19.5)

14. Primary Outcome: First Order Elimination Rate Constant Associated With the Terminal (Log-linear) Portion of the Curve (Lambda z) of Lanadelumab
Description: Lambda z of Lanadelumab was reported.
Time Frame: Pre-dose (Day 1) up to 2664 hours post-dose
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Per hour (/h)
Arm/Group | Lanadelumab 300 mg
Number analyzed (Participants) | 9
Per hour (/h) | 9.90 (31.0)

ADVERSE EVENTS:
Time Frame: From the first dose of study treatment up to the end of study (Day 112)
Arm/Group | Lanadelumab 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/3
Other Adverse Events (participants affected / at risk) | 7/9 | 2/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lanadelumab 300 mg (N=9) | Placebo (N=3)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 2 (4) | 1 (2)
Paraesthesia (Nervous system disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.

DOCUMENTS (2):
  • Study Protocol (2020-09-16): https://cdn.clinicaltrials.gov/large-docs/03/NCT04503603/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/03/NCT04503603/SAP_001.pdf